CLINICAL TRIAL: NCT00122616
Title: Efficacy of Pegylated Interferon on Liver Fibrosis in Co-infected Patient With HIV and C Hepatitis Who Failed to Active Treatment for HCV. ANRSHC12 Fibrostop
Brief Title: Efficacy of Pegylated Interferon on Liver Fibrosis in Co-infected Patient With HIV and Hepatitis C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRSHC12 FIBROSTOP
Record Dates: First submitted 2005-07-19; First posted 2005-07-22 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: HIV Infections; Hepatitis C, Chronic
Keywords: HIV infections; peginterferon alfa-2a; Treatment Failure; Hepatitis C, Chronic; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peginterféron alpha-2a + Ribavirin+ HIV antiretroviral therapy (Active Comparator): Day0 to week 96:Peginterféron alpha-2a + Ribavirin+ HIV antiretroviral therapy
  Interventions: Biological: Peginterferon alpha-2a (Pegasys®); Drug: Ribavirin; Drug: HIV antiretroviral therapy
- HIV antiretroviral therapy (Placebo Comparator): Day0 to week 96: HIV antiretroviral therapy
  Interventions: Drug: HIV antiretroviral therapy

INTERVENTIONS:
Biological: Peginterferon alpha-2a (Pegasys®) — Peg-Interferon Alpha2a by subcutaneous injection, 180µg, once weekly
  Arms: Peginterféron alpha-2a + Ribavirin+ HIV antiretroviral therapy
Drug: Ribavirin — Ribavirin: tablet oral, weight-based dose, 1000 mg for subjects weighing below 75 kg or 1200 mg for subjects weighing equal or over 75 kg, once daily
  Arms: Peginterféron alpha-2a + Ribavirin+ HIV antiretroviral therapy
Drug: HIV antiretroviral therapy — All antiretroviral drugs are allowed, their choice being left to the discretion of the investigator. Particular attention will be carried to the patients with antiretroviral susceptible to cause a cumulative toxicity with anti-VHC drugs
  Arms: Peginterféron alpha-2a + Ribavirin+ HIV antiretroviral therapy
Drug: HIV antiretroviral therapy — All antiretroviral drugs are allowed, their choice being left to the discretion of the investigator. Particular attention will be carried to the patients with antiretroviral susceptible to cause a cumulative toxicity with anti-VHC drugs
  Arms: HIV antiretroviral therapy

SUMMARY:
The aim of this study is to prove the efficacy of peginterferon in HIV infected patients with liver disease caused by hepatitis C virus (HCV) when the treatment to eradicate the virus failed. This scientific proof needs a comparative study to be done including two groups of patients randomly allocated: one with the treatment (peginterferon) and the other without any treatment against HCV with a duration of 2 years. To conclude, two liver biopsies are needed; one before the study and a second 2 years after.

DETAILED DESCRIPTION:
C hepatitis in HIV infected patient becomes a major issue although the survival of patients, has improved in the last decades regarding to the advent of HAART, the mortality related to liver disease has increased in this population. Sustained virological response for HCV can be obtained with peg-interferon and ribavirin treatment but more or less 50% of patients experienced failure to this treatment and liver fibrosis due to HCV infection progress and may lead to cirrhosis and hepato-carcinoma. To demonstrate the efficacy of peginterferon therapy to reduce the liver damage causes by HCV infection, a randomised controlled study is needed comparing one group of patient treated by peginterferon and one group without any treatment against HCV infection. In order to show 30% difference between the two groups in reducing one point of fibrosis score (METAVIR scale), 150 patients are needed. The duration of the study is 96 weeks

ELIGIBILITY:
Inclusion Criteria:

* HIV infection (Western Blot +)
* C hepatitis (RNA viral hepatitis C [VHC] +)
* Chronic active C hepatitis on liver histological score METAVIR (A over or equal to 1 and F over or equal to 2) on biopsy performed at least 18 months before the expected date of inclusion
* Previous treatment for C hepatitis for at least 3 months including peg-interferon and ribavirin or peg-interferon alone if counterindication for ribavirin occurred
* Failure to eradicate C hepatitis virus after well conducted treatment
* The liver biopsy should have been realised at least 18 months before inclusion :

Either before treatment for C hepatitis in patients treated at most 7 months Or at least 6 months after anti HCV treatment in patient treated for more than 7 months (wash out period)

* Regular follow up in an outpatient clinic for HIV
* Unchanged antiretroviral treatment the last 3 months before inclusion
* Inform consent

Exclusion Criteria:

* History of transplantation or clinical hepatic failure
* Opportunistic infection in the past three months before inclusion
* Any hepatic disease not related to HCV (B hepatitis, hemochromatosis, Wilson disease)
* Diabetes mellitus
* Immunocompromised treatment
* Active intravenous drug addiction
* Alcohol consumption of more than 50 g per day
* Counterindication for the use of interferon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2003-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who experienced one point decreases of their fibrosis histological score (Metavir). | Week 96

SECONDARY OUTCOMES:
Distribution of the change of fibrosis Metavir score in each group | Week 96
Distribution of fibrosis score from Chevallier classification | Week 96
Plasmatic fibrosis markers dosages | Week 96
Viral load quantification for HIV and HCV | Week 96
Number and percentage of CD4/CD8 cell count throughout the study | Day 0 to week 96
Number and percentage of patient had more thand 200 copies/ml throughout the study | Day 0 to week 96
Occurrence of hepatic complication related to HCV | Day0 to week 96
Survival throughout the study | Day 0 to week 96
Quality of life questionnaire | Day 0 to week 96
Fibrotest (plasmatic fibrosis marker) | Day 0, week 48 and week 96
Histological improvement according to the total interferon dose received | Day 0 to week 96

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marc Chapplain, MD, Principal Investigator — Hopital Pontchaillou Rennes; Eric Belissant, MD, Study Chair — CIC Hôpital Pontchaillou Rennes
Locations (1):
- Service de Maladies Infectieuses et de Réanimation Médicale, Rennes, France

REFERENCES:
- [Derived] Chapplain JM, Bellissant E, Guyader D, Molina JM, Poizot-Martin I, Perre P, Pialoux G, Turlin B, Mouchel C, Renault A, Michelet C; ANRS HC-12 Study Group. The effects of a maintenance therapy with peg-interferon alpha-2a on liver fibrosis in HIV/HCV co-infected patients: a randomized controlled trial. J Infect. 2013 Oct;67(4):313-21. doi: 10.1016/j.jinf.2013.05.007. Epub 2013 Jun 22. PMID 23800784